CLINICAL TRIAL: NCT05687331
Title: Changes in the Immunomodulatory Properties of Adipose Stromal Cells Due to Hemarthrosis After Knee Injury
Acronym: CASH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL77974.091.21
Record Dates: First submitted 2022-12-13; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Post-Traumatic Osteoarthritis of Knee; Knee Injuries; Hemarthrosis
MeSH Terms: conditions — Knee Injuries; Hemarthrosis | interventions — Phlebotomy; Blood Specimen Collection; Magnetic Resonance Imaging; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma, synovial fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hemarthrosis: 10 patients that sustained a knee trauma and have hemarthrosis during knee arthrocentesis (red color of the synovial fluid)
  Interventions: Procedure: knee arthrocentesis; Procedure: venipuncture; Diagnostic Test: MRI-scan; Diagnostic Test: Physical examination; Other: KOOS questionnaire
- Patients without hemarthrosis: 10 patients that sustained a knee trauma and do not have hemarthrosis during knee arthrocentesis (yellow color of the synovial fluid)
  Interventions: Procedure: knee arthrocentesis; Procedure: venipuncture; Diagnostic Test: MRI-scan; Diagnostic Test: Physical examination; Other: KOOS questionnaire

INTERVENTIONS:
Procedure: knee arthrocentesis — arthrocentesis of the knee joint to gather a synovial fluid sample
Procedure: venipuncture — Peripheral venipuncture to gather a blood sample
  Other Names: blood draw
Diagnostic Test: MRI-scan — MRI-scan of the knee
Diagnostic Test: Physical examination — Physical examination of the injured knee
Other: KOOS questionnaire — KOOS questionnaire of the injured knee

SUMMARY:
The goal of this observational study is to gain insight in the natural course of pro-inflammatory factors and hemarthrosis in patients older than 18 with a recent knee trauma. The main question[s] it aims to answer are:

* What is the natural course of pro-inflammatory factors and hemarthrosis in knee trauma?
* What are the effects of inflammation and hemarthrosis on the anti-inflammatory potential of ASC's in order to better determine eligible patients and circumstances for ASC's therapy?

Participants will:

* undergo blood withdrawal
* undergo knee arthrocentesis for synovial fluid sample collection
* physical examination
* fill out a questionnaire on knee complaints

DETAILED DESCRIPTION:
Recent studies have found an amelioration of post-traumatic osteoarthritis by the use of adipose-derived stromal cells (ASC's) in an experimental animal model. This amelioration was only seen under inflammatory conditions. The presence of hemarthrosis has not been taken into account in the before mentioned animal model, and might have cytotoxic effects on ASC's and aggravate the inflammatory response. The objective of this study is to gain insight in the natural course of pro-inflammatory factors and hemarthrosis and its effects on the anti-inflammatory potential of ASC's in order to better determine eligible patients and circumstances for ASC's therapy.

Therefore the investigators designed a pilot study with exploratory analyses in and with synovial fluid in a longitudinal cohort.

Our study population will consist of 20 patients, older than 18 years, who sustained a recent knee trauma and are presented to the emergency department.The investigators will gather synovial fluid and blood samples for laboratory analysis perform and physical examination and provide questionnaires for clinical follow-up.

The main study endpoint are the anti-inflammatory capacities of ASC's in synovial fluid that contains blood as a result of hemarthrosis after knee injury.

ELIGIBILITY:
Inclusion Criteria:

* Recently suffered an injury of the index knee (rotational or hyperextension)
* A swollen joint
* Inability to mobilise

Exclusion Criteria:

* Patients with an active inflammatory or infectious comorbid disease (including rheumatic diseases)
* Patients using systemic immunosuppressant medication
* Patients with a contra-indication for undergoing a MRI-scan (non-compatible implants or claustrophobia for example)
* Patients with knee prosthesis
* Patients with coagulation disorders
* Patients with a history of a cruciate ligament or meniscal injury of the index knee
* Patients with a tibiofemoral fracture of the index knee due to current distortion
* In case the inclusion of the required amount of patient is reached in one the patient groups, additional patients belonging in the same patient group will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who are presented at the emergency department of the CWZ hospital because of a recent distortion of the knee.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Synovial fluid analysis | Samples are taken at week 1, week 2, week 4, week 6 and week 8 after trauma
  Analysis of changes in pro-inflammatory factors, erythrocytes (as measurement for hemarthrosis)

SECONDARY OUTCOMES:
co-culture of synovial fluid with adipose stromal cells | samples are taken at week 1, week 2, week 4, week 6 and week 8 after trauma
  Assessment of changes in cytotoxity of hemarthrosis in synovial fluid on adipose stromal cells
MRI-imaging | At inclusion and 1 year after trauma
  MRI-images to determine post-traumatic changes in the articulate cartilage
Physical examination | Physical examination at week 1, week 2, week 4, week 6 and week 8 after trauma
  Assessment of changes in swelling, warmth and appearance of the skin
Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire | Questionnaires are taken at week 1, week 2, week 4, week 6 and week 8 after trauma
  Assessment changes of knee complaints by using the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire, with minimum score of 0 and a maximum score of 100 and a higher score meaning a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud umc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Riordan EA, Little C, Hunter D. Pathogenesis of post-traumatic OA with a view to intervention. Best Pract Res Clin Rheumatol. 2014 Feb;28(1):17-30. doi: 10.1016/j.berh.2014.02.001. PMID 24792943
- [Background] Lohmander LS, Englund PM, Dahl LL, Roos EM. The long-term consequence of anterior cruciate ligament and meniscus injuries: osteoarthritis. Am J Sports Med. 2007 Oct;35(10):1756-69. doi: 10.1177/0363546507307396. Epub 2007 Aug 29. PMID 17761605
- [Background] Luc B, Gribble PA, Pietrosimone BG. Osteoarthritis prevalence following anterior cruciate ligament reconstruction: a systematic review and numbers-needed-to-treat analysis. J Athl Train. 2014 Nov-Dec;49(6):806-19. doi: 10.4085/1062-6050-49.3.35. PMID 25232663
- [Background] Ayral X, Pickering EH, Woodworth TG, Mackillop N, Dougados M. Synovitis: a potential predictive factor of structural progression of medial tibiofemoral knee osteoarthritis -- results of a 1 year longitudinal arthroscopic study in 422 patients. Osteoarthritis Cartilage. 2005 May;13(5):361-7. doi: 10.1016/j.joca.2005.01.005. PMID 15882559
- [Background] Pulles AE, Mastbergen SC, Schutgens RE, Lafeber FP, van Vulpen LF. Pathophysiology of hemophilic arthropathy and potential targets for therapy. Pharmacol Res. 2017 Jan;115:192-199. doi: 10.1016/j.phrs.2016.11.032. Epub 2016 Nov 24. PMID 27890816
- [Background] Gupte C, St Mart JP. The acute swollen knee: diagnosis and management. J R Soc Med. 2013 Jul;106(7):259-68. doi: 10.1177/0141076813482831. PMID 23821708
- [Background] Wang Y, Shimmin A, Ghosh P, Marks P, Linklater J, Connell D, Hall S, Skerrett D, Itescu S, Cicuttini FM. Safety, tolerability, clinical, and joint structural outcomes of a single intra-articular injection of allogeneic mesenchymal precursor cells in patients following anterior cruciate ligament reconstruction: a controlled double-blind randomised trial. Arthritis Res Ther. 2017 Aug 2;19(1):180. doi: 10.1186/s13075-017-1391-0. PMID 28768528
- [Background] ter Huurne M, Schelbergen R, Blattes R, Blom A, de Munter W, Grevers LC, Jeanson J, Noel D, Casteilla L, Jorgensen C, van den Berg W, van Lent PL. Antiinflammatory and chondroprotective effects of intraarticular injection of adipose-derived stem cells in experimental osteoarthritis. Arthritis Rheum. 2012 Nov;64(11):3604-13. doi: 10.1002/art.34626. PMID 22961401
- [Background] Schelbergen RF, van Dalen S, ter Huurne M, Roth J, Vogl T, Noel D, Jorgensen C, van den Berg WB, van de Loo FA, Blom AB, van Lent PL. Treatment efficacy of adipose-derived stem cells in experimental osteoarthritis is driven by high synovial activation and reflected by S100A8/A9 serum levels. Osteoarthritis Cartilage. 2014 Aug;22(8):1158-66. doi: 10.1016/j.joca.2014.05.022. Epub 2014 Jun 10. PMID 24928317
- [Background] Pers YM, Rackwitz L, Ferreira R, Pullig O, Delfour C, Barry F, Sensebe L, Casteilla L, Fleury S, Bourin P, Noel D, Canovas F, Cyteval C, Lisignoli G, Schrauth J, Haddad D, Domergue S, Noeth U, Jorgensen C; ADIPOA Consortium. Adipose Mesenchymal Stromal Cell-Based Therapy for Severe Osteoarthritis of the Knee: A Phase I Dose-Escalation Trial. Stem Cells Transl Med. 2016 Jul;5(7):847-56. doi: 10.5966/sctm.2015-0245. Epub 2016 May 23. PMID 27217345